CLINICAL TRIAL: NCT03542877
Title: An Open-Label, Single-Arm, Two-Stage Phase II Study Investigating Cabozantinib in Patients With Refractory Metastatic Colorectal Cancer
Brief Title: Investigating Cabozantinib in Patients With Refractory Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic Thoracic Oncology Medical Investigators Consortium (Industry)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Organization: University of Colorado, Denver (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0021.cc
Record Dates: First submitted 2018-04-23; First posted 2018-05-31 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer
Keywords: Cabozantinib; Progression Free Survival; Metastatic Colorectal Cancer; Tumor
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Cabozantinib (Experimental): Patients will be enrolled to take 60mg of cabozantinib, by mouth, once a day, every day, for 12 weeks. If less than three patients have Progression Free Survival (PFS) lasting at least 12 weeks, the study will be terminated.
  Interventions: Drug: Oral Tablet: Cabozantinib

INTERVENTIONS:
Drug: Oral Tablet: Cabozantinib — Patients will take 60mg cabozantinib, by mouth, once daily, every day for 12 weeks. This medication should be taken on an empty stomach. Patients should not eat 2 hours before or 1 hour after taking cabozantinib. Only water is permitted during this 3 hour time frame.
  Other Names: Cometriq; Cabometyx

SUMMARY:
This study seeks to use Cabozantinib to treat those with Metastatic Colorectal Cancer who have not previously responded to treatment.

DETAILED DESCRIPTION:
This is a phase II clinical trial that seeks to use Cabozantinib to treat those with Metastatic Colorectal Cancer who have not previously responded to treatment. This study is a two stage study that will first measure (up to) 16 patients' progression free survival (PFS). Stage two will, again, measure PFS, but in a population (up to) 28 patients.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a histologic or cytologic diagnosis of colorectal adenocarcinoma that is metastatic or unresectable and is refractory to or progressed (or relapsed) following a fluoropyrimidine, irinotecan, oxaliplatin, and bevacizumab; prior epidermal growth factor inhibitor therapy is required for patients with left-sided, RAS wild-type tumors; prior FDA-approved PD-1 inhibitor therapy is required for patients with MSI-H colorectal cancer. Prior regorafenib or TAS-102 treatment is not required.
2. Measurable disease per RECIST 1.1 as determined by the investigator.
3. The subject has had an assessment of all known disease sites e.g., by computerized tomography (CT) scan and/or magnetic resonance imaging (MRI) within 28 days before the first dose of cabozantinib.
4. The subject is ≥ 18 years old on the day of consent.
5. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Recovery to baseline or ≤ Grade 1 CTCAE v.4.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
7. Adequate archival frozen or fixed tissue available from primary or metastatic site for genotypic analysis (at least 15 unstained slides and/or tumor block).
8. The subject has organ and marrow function and laboratory values as follows within 7 days before the first dose of cabozantinib:

   1. ANC ≥ 1500/mm3 without colony stimulating factor support;
   2. Platelets ≥ 100,000/mm3;
   3. Hemoglobin ≥ 9 g/dL;
   4. Bilirubin ≤ 1.5 x ULN. For subjects with known Gilbert's disease, bilirubin ≤ 3.0 mg/dL;
   5. Serum albumin ≥ 2.8 g/dl;
   6. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used:

      * Male: CrCl (mL/min) = (140 - age) × wt (kg) / (serum creatinine × 72);
      * Female: Multiply above result by 0.85;
   7. ALT and AST ≤ 3.0 x ULN;
   8. Lipase < 2.0 x the upper limit of normal and no radiologic or clinical evidence of pancreatitis;
   9. UPCR ≤ 1;
   10. Serum phosphorus, calcium, magnesium and potassium ≥ LLN.
9. The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.
10. Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control or practice abstinence during the study and for 4 months after the last dose of study drug(s).

Exclusion Criteria:

1. The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (eg, cytokines or antibodies) within 3 weeks, or nitrosoureas/mitomycin C within 6 weeks before the first dose of study treatment;
2. Prior treatment with cabozantinib;
3. Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before the first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible;
4. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 14 days before the first dose of study treatment. Note: Subjects with prostate cancer currently receiving LHRH or GnRH agonists may be maintained on these agents;
5. The subject has received any other type of investigational agent within 28 days before the first dose of study treatment;
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before the first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the start of study treatment;
7. The subject has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.3 x the laboratory ULN within 7 days before the first dose of study treatment;
8. Concomitant anticoagulation at therapeutic doses with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel); Note: Low-dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (< 1 mg/day), and low dose, low molecular weight heparins (LMWH) are permitted. Anticoagulation with therapeutic doses of LMWH is allowed in subjects without radiographic evidence of brain metastasis, who are on a stable dose of LMWH for at least 12 weeks before randomization, and who have had no complications from a thromboembolic event or the anticoagulation regimen. ;
9. The subject has experienced any of the following:

   1. clinically-significant GI bleeding within 6 months before the first dose of study treatment;
   2. hemoptysis of ≥ 0.5 teaspoon (2.5ml) of red blood within 3 months before the first dose of study treatment;
   3. any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment.
10. The subject has radiographic evidence of cavitating pulmonary lesion(s);
11. The subject has tumor invading or encasing any major blood vessels;
12. The subject has evidence of clinically significant bleeding from tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib;
13. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

    a. Cardiovascular disorders including: i. Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening; ii. Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment; iii. Any history of congenital long QT syndrome; iv. Any of the following within 6 months before the first dose of study treatment:
    * unstable angina pectoris;
    * clinically-significant cardiac arrhythmias;
    * stroke (including transient ischemic attack (TIA), or other ischemic event);
    * myocardial infarction;
    * thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (eg, vena cava filter) are not eligible for this study).

      b. GI disorders particularly those associated with a high risk of perforation or fistula formation including: i. Active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction ii. Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before randomization, Note: Complete healing of an intra-abdominal abscess must be confirmed prior to randomization c. Other clinically significant disorders that would preclude safe study participation;
14. Major surgery within 12 weeks before the first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment. Minor surgery (including uncomplicated tooth extractions) within 28 days before the first dose of study treatment with complete wound healing at least 10 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible;
15. QTcF > 500 msec within 1 month before the first dose of study treatment:

    a. Three ECGs must be performed for eligibility determination. If the average of these three consecutive results for QTcF is ≤ 500 msec, the subject meets eligibility in this regard.
16. Pregnant or lactating females;
17. Inability to swallow intact tablets;
18. Previously identified allergy or hypersensitivity to components of the study treatment formulations;
19. Diagnosis of another malignancy within 2 years before the first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, MD, Principal Investigator — University of Colorado, Denver
Locations (10):
- United States (10):
  - University of Arizona, Tucson, Arizona
  - Kenneth Norris Jr. Comprehensive Cancer Center, Los Angeles, California
  - Universtiy of Colorado Denver, Aurora, Colorado
  - Lone Tree Health Center, Lone Tree, Colorado
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Swedish Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Cabozantinib
Started | 44
Completed | 23
Not Completed | 21

BASELINE CHARACTERISTICS:
Arm/Group | Oral Cabozantinib
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (23)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 13
  Male | 30
  Unknown | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 38
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: 12-Week Progression Free Survival
Description: A patient is classified as progression-free if s/he is assessed as not having progressive disease (PD) as defined per RECIST 1.1 criteria at either the 12-week assessment or after having at least 11 weeks of treatment for subjects without the 12-week assessment. Censored patients (i.e. those who have not progressed but who are missing a 12-week assessment) are not included in the analysis. Subjects who didn't have the 12-week assessment but who had clinical progression were included and considered to have progressed.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECISTv1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: This outcome was assessed at the 12-week assessment. Subjects without the 12-week assessment but who had at least 11 weeks of treatment were included.
Population: 40 of the 44 subjects were in the analysis population. 3 subjects were not included because they didn't have treatment response data, and 1 subject was not included because that subject didn't reach at least week 11 (and didn't have PD).
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Cabozantinib
Number analyzed (Participants) | 40
Participants | 18

2. Secondary Outcome: 12-Week Progression-Free Survival by RAS Mutation Status
Description: This has the same outcome measure description as the primary analysis. Per Response Evaluation Criteria In Solid Tumors Criteria (RECISTv1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: as for outcome 1
Population: This population was the same as the population for the primary analysis
Measure: Count of Participants; unit: Participants
Groups:
- RAS Mutant: Subjects who were RAS mutant.
- RAS Wild Type: Subjects with wild type RAS mutation status
Arm/Group | RAS Mutant | RAS Wild Type
Number analyzed (Participants) | 22 | 18
Participants | 7 | 11

3. Secondary Outcome: 12-Week Progression-Free Survival by PIK3CA Mutation Status
Description: as for outcome 2
Time Frame: as for outcome 1
Population: All subjects in the primary analysis who had data regarding their PIK3CA mutation status.
Measure: Count of Participants; unit: Participants
Groups:
- PIK3CA Mutant: Subjects who were PIK3CA mutant.
- PIK3CA Wild Type: Subjects with wild type PIK3CA mutation status.
Arm/Group | PIK3CA Mutant | PIK3CA Wild Type
Number analyzed (Participants) | 6 | 22
Participants | 3 | 11

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival will be defined as the time from administration of the initial dose of cabozantinib to evidence of radiographic progression as defined by RECIST criteria or death from any cause without evidence of disease progression, whichever occurs first.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECISTv1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Study start date to study end date, or death, whichever comes first, up to 24 months
Population: 3 of the 44 study subjects were not included in this analysis population because they didn't have treatment response data.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Oral Cabozantinib
Number analyzed (Participants) | 41
Weeks | 13 [9 to 21]

5. Secondary Outcome: Progression-Free Survival (PFS) by RAS Mutation Status
Description: This has the same outcome measure description as the PFS analysis. Per Response Evaluation Criteria In Solid Tumors Criteria (RECISTv1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Study start date to study end date, or death, whichever comes first, up to 24 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | RAS Mutant | RAS Wild Type
Number analyzed (Participants) | 23 | 18
Weeks | 12 [6 to 14] | 21 [9 to 48]

6. Secondary Outcome: Progression-Free Survival (PFS) by PIK3CA Mutation Status
Description: as for outcome 5
Time Frame: Study start date to study end date, or death, whichever comes first, up to 24 months
Population: All subjects in the PFS secondary analysis who had data regarding their PIK3CA mutation status.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | PIK3CA Mutant | PIK3CA Wild Type
Number analyzed (Participants) | 7 | 22
Weeks | 26 [5 to NA] — The upper limit of this 95% CI is infinity (and the entry 'Infinity' cannot be made) | 20 [6 to 29]

7. Secondary Outcome: Response Rate in Patients With CRC Treated With Cabozantinib
Description: *A patient is classified as a responder if s/he is assessed as having complete response or partial response (CR or PR) at the time of any assessment, where CR and PR are defined per RECIST 1.1 criteria.
Time Frame: Study start date to study end date, or death, whichever comes first, up to 24 months
Population: This analysis population was the same as described for the primary analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Cabozantinib
Number analyzed (Participants) | 40
Participants | 1

8. Secondary Outcome: Overall Survival (OS) in Patients With CRC Treated With Cabozantinib
Description: Overall Survival will be defined as the time from administration of the initial dose of cabozantinib until death from any cause.
Time Frame: Study start date to study end date, or death, whichever comes first, up to 24 months
Population: All 34 subjects with follow-up data (i.e. data in the 'dataset_survival_follow_up.xlsx' table) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Oral Cabozantinib
Number analyzed (Participants) | 34
Weeks | 36 [24 to 50]

9. Secondary Outcome: Overall Survival (OS) by RAS Mutation Status
Description: This has the same outcome measure description as the OS analysis.
Time Frame: Study start date to study end date, or death, whichever comes first, up to 24 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | RAS Mutant | RAS Wild Type
Number analyzed (Participants) | 19 | 15
Weeks | 30 [18 to 46] | 45 [20 to NA] — The upper limit of the 95% CI is Infinity (which isn't an acceptable entry above)

10. Secondary Outcome: Overall Survival (OS) by PIK3CA Mutation Status
Description: This has the same outcome measure description as the OS analysis.
Time Frame: Study start date to study end date, or death, whichever comes first, up to 24 months
Population: All subjects in the secondary OS analysis who had data regarding their PIK3CA mutation status.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | PIK3CA Mutant | PIK3CA Wild Type
Number analyzed (Participants) | 5 | 17
Weeks | 92 [9 to NA] — The upper limit of the 95% CI is Infinity (which is not an acceptable entry above) | 36 [20 to 85]

ADVERSE EVENTS:
Time Frame: 45 months
Arm/Group | Oral Cabozantinib
All-Cause Mortality (participants affected / at risk) | 5/44
Serious Adverse Events (participants affected / at risk) | 20/44
Other Adverse Events (participants affected / at risk) | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Cabozantinib (N=44)
Cavitating Pulmonary Nodules (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Acute Cerebrovascular Accident (General disorders) | 1 (1)
Acute Pancreatitis (Gastrointestinal disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Back Pain (General disorders) | 1 (1)
Bowel Perforation (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Dehydration (General disorders) | 1 (1)
difficulty speaking (General disorders) | 1 (1)
Disease Progression (General disorders) | 2 (2)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1)
Duodenal fistula (Gastrointestinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Failure to Thrive (General disorders) | 1 (1)
GI bleed (Gastrointestinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 1 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Progressed Malignant Neoplasm (General disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Severe Complicated Bilateral Pyelonephritis (Renal and urinary disorders) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Cabozantinib (N=44)
Abdominal Pain (Gastrointestinal disorders) | 16 (19)
Abdominal Distension (Gastrointestinal disorders) | 1 (2)
Acid Reflux (Gastrointestinal disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 3 (3)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 2 (2)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 7 (8)
Alopecia (General disorders) | 3 (3)
alanine aminotransferase increase (Blood and lymphatic system disorders) | 7 (10)
Amylase increased (Blood and lymphatic system disorders) | 3 (4)
Anemia (Blood and lymphatic system disorders) | 7 (8)
Anorexia (General disorders) | 16 (26)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 9 (19)
Hearing Loss (General disorders) | 1 (1)
Edema (Blood and lymphatic system disorders) | 9 (12)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 12 (20)
Hypertension (Blood and lymphatic system disorders) | 15 (31)
Mouth Sores (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (General disorders) | 17 (19)
Elevated Creatinine (Blood and lymphatic system disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 14 (15)
Diarrhea (Gastrointestinal disorders) | 23 (33)
Hypokalemia (Blood and lymphatic system disorders) | 8 (11)
Mouth Sensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Skin sensitivity (Skin and subcutaneous tissue disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 10 (11)
Rash (Skin and subcutaneous tissue disorders) | 6 (9)
sinusitis (General disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 12 (17)
Fatigue (General disorders) | 28 (48)
chest pain (General disorders) | 3 (3)
thrombocytopenia (Blood and lymphatic system disorders) | 8 (9)
Elevated troponin (Cardiac disorders) | 1 (1)
fecal impaction (Gastrointestinal disorders) | 1 (1)
sore throat (General disorders) | 6 (7)
Cramping (Musculoskeletal and connective tissue disorders) | 10 (11)
hoarse (General disorders) | 4 (4)
palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 14 (35)
Chills (General disorders) | 4 (4)
fever (General disorders) | 8 (9)
forgetfulness (General disorders) | 3 (3)
Reflux (Gastrointestinal disorders) | 9 (9)
Elevated Liver Function Test (Blood and lymphatic system disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Mucositis (Skin and subcutaneous tissue disorders) | 5 (5)
Neuropathy (Nervous system disorders) | 7 (7)
Tachycardia (Cardiac disorders) | 1 (1)
Lactate Increased (Blood and lymphatic system disorders) | 1 (1)
Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Tenderness (General disorders) | 1 (1)
Pain (General disorders) | 17 (38)
Ache (General disorders) | 6 (9)
Distended Abdomen (Gastrointestinal disorders) | 2 (3)
Weakness (General disorders) | 2 (2)
Xerostomia (Skin and subcutaneous tissue disorders) | 4 (4)
Hyperamylasemia (Blood and lymphatic system disorders) | 5 (7)
Decreased Appetite (General disorders) | 2 (2)
Congestion (General disorders) | 3 (4)
Bleeding gums (General disorders) | 1 (1)
Malnutrition (General disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 14 (19)
Dizziness (General disorders) | 7 (9)
Dysgeusia (General disorders) | 7 (7)
Cough (General disorders) | 7 (9)
Infection (Infections and infestations) | 1 (1)
Hematuria (Renal and urinary disorders) | 7 (10)
TSH elevated (Endocrine disorders) | 4 (4)
epistaxis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (3)
Bilirubin Increased (Blood and lymphatic system disorders) | 6 (12)
bradycardia (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Gait Disturbance (General disorders) | 2 (2)
Dysesthesia (General disorders) | 2 (2)
Hypersomnia (General disorders) | 1 (1)
Blurred vision (General disorders) | 3 (3)
Weight Gain (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Renal and urinary disorders) | 1 (1)
Conduction Disorder (Cardiac disorders) | 1 (1)
hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Dental Caries (General disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hyperlipasemia (Blood and lymphatic system disorders) | 4 (5)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 2 (2)
Lymphocytopenia (Blood and lymphatic system disorders) | 3 (3)
Hyperglycemia (Endocrine disorders) | 3 (4)
Hypernatremia (Blood and lymphatic system disorders) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 4 (4)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 6 (9)
Ascites (Blood and lymphatic system disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3)
Tonsilitis (Infections and infestations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Mood alteration (Psychiatric disorders) | 2 (2)
Hypertention (Vascular disorders) | 3 (8)
Numbness of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Elevated Urine Protein Creatinine Ratio (Renal and urinary disorders) | 2 (4)
Increased Creatinine (Renal and urinary disorders) | 1 (1)
Migraine (General disorders) | 2 (2)
Change in Hair Color (General disorders) | 2 (3)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Burning mouth syndrom (Skin and subcutaneous tissue disorders) | 1 (1)
Wound bleeding (Injury, poisoning and procedural complications) | 1 (1)
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Urine Discoloration (Renal and urinary disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Pancreatitis (Infections and infestations) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Neurological Changes (General disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Tumor Lysis Syndrome (Blood and lymphatic system disorders) | 1 (1)
Diaphoresis (General disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 2 (2)
Laryngitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT03542877/Prot_SAP_000.pdf